CLINICAL TRIAL: NCT05063279
Title: Resistance Training for Life - the Efficacy of Increasing Resistance Training Volume for Improving Muscle Mass, Function, Biology and Health in Young and Elderly
Brief Title: RELIEF - Resistance Training for Life
Acronym: RELIEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stian Ellefsen (Other)
Collaborators: Sykehuset Innlandet HF (Other)
Responsible Party: Sponsor-Investigator, Stian Ellefsen, Professor, Inland Norway University of Applied Sciences
Organization: Inland Norway University of Applied Sciences (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: TR030
Record Dates: First submitted 2021-09-11; First posted 2021-10-01 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: Study conditions (exercise volume) are randomized to either leg/arm for within-participant comparisons. The effect of age is assessed from two parallel age groups.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Study conditions (exercise volume) and age groups identifiers are omitted from outcome assessments whenever possible. Assessment of the primary (and selected secondary) outcome(s) will be performed in a blinded fashion by assessors/investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance training group (Experimental): Participants in two age groups will receive moderate (three sets of per exercise per session) and low-volume (one set of resistance per session) training allocated to either right or left upper- and lower extremities. A total of 24 sessions will be performed over 10-12 weeks.
  Interventions: Other: Progressive resistance training
- Negative control group (No Intervention): A negative control group is included in the study which will not receive any resistance training.

INTERVENTIONS:
Other: Progressive resistance training — Progressive resistance training, performed with a target number of repetitions of 10 per set. Sets are performed to exhaustion, and external load will be adjusted to meet the target number of repetitions.
  Arms: Resistance training group

SUMMARY:
Sarcopenia is an age-related gradual loss of muscle mass and strength and is associated with physical disability and mortality risk. Currently, the most promising remedy for preventing and treating sarcopenia is physical activity, particularly progressive resistance training. Yet, the amount of resistance exercise needed to achieve optimal benefits remains largely unknown. This lack of knowledge is underpinned by the notion that aging reduces the ability to adapt to (and benefit from) resistance training, and is further complicated by a relative large degrees of between-subject heterogeneity. The primary aim of the study is to compare the effects of 10 weeks of resistance training with low- and moderate volume (one vs. three sets per exercise) on muscle mass accretion in lower and upper body extremities in young (<30 years of age) and elderly individuals (>70 years of age). Specifically, the study addresses the hypothesis that elderly individuals will benefit more from higher exercise volume (moderate vs. low) compared to their young counterparts. In addition, the study aims to compare the efficacy of the two volume conditions for altering other characteristics such as muscle strength and biology, including assessment of associations between individual changes in muscle mass, strength and biology (e.g. the relationship between muscle mass accretion and muscle content of rRNA/rDNA), and also to investigate the general health effects of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18 and 30 or > 70

Exclusion Criteria:

* Resistance training, > 1 session per week
* Endurance training, > 3 sessions per week
* Unstable cardiovascular disease
* Illness or serious injury contradicting resistance training
* Serious mental illness
* Allergy to local anaesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Muscle size, lower extremities | Change from baseline to after the training period (10-12 weeks)
  Muscle size of lower extremity knee extensors measured with magnetic resonance imaging (MRI).

SECONDARY OUTCOMES:
Muscle size, upper-body extremities | Change from baseline to after the training period (10-12 weeks)
  Muscle size of upper extremity elbow flexors measured with magnetic resonance imaging (MRI).
Appendicular lean mass, lower-body extremities | Change from baseline to after the training period (10-12 weeks)
  Appendicular lean mass of the legs measured using Dual X-Ray Absorptiometry
Appendicular lean mass, upper-body extremities | Change from baseline to after the training period (10-12 weeks)
  Appendicular lean mass of the arms measured using Dual X-Ray Absorptiometry
Muscle thickness, m. vastus lateralis | Change from baseline to after the training period (10-12 weeks)
  Musle thickness of m. vastus lateralis measured using ultrasound
Muscle strength, lower-body extremities | Change from baseline to after the training period (10-12 weeks)
  Muscle strength of the legs measured as a weighted average of lower body isokinetic and isometric knee extensor maximal force
Muscle strength, upper-body extremities | Change from baseline to after the training period (10-12 weeks)
  Muscle strength of the arms measured as isometric force (elbow flexors; fixed angle)
Muscular peak power/force, lower-body extremities | MeasurChange from baseline to after the training period (10-12 weeks)
  Muscular peak power/force measured using dynamic leg press

OTHER OUTCOMES:
Muscle thickness, m. vastus lateralis (mid) | Change from baseline to after 12 sessions
  Musle thickness of m. vastus lateralis measured using ultrasound
Muscle strength, lower-body extremities (mid) | Change from baseline to after 12 sessions
  Muscle strength will be assessed as a weighted average of lower body isokinetic and isometric knee extensor maximal force
Muscle strength, upper-body extremities (mid) | Change from baseline to after 12 sessions
  Muscle strength of the arms measured as isometric force (elbow flexors; fixed angle)
Muscular peak power/force, lower-body extremities | Change from baseline to after 12 sessions
  Muscular peak power/force measured using dynamic leg press
Muscle architecture, m. vastus lateralis (mid) | Change from baseline to after 12 sessions
  Muscle architecture pennation angle of m. vastus lateralis measured using ultrasound
Muscle architecture, m. vastus lateralis | Change from baseline to the training period (10-12 weeks).
  Muscle architecture pennation angle of m. vastus lateralis measured using ultrasound
Body composition | Change from baseline to after the training period (10-12 weeks).
  Whole Body Dual X-Ray Absorptiometry to estimate lean mass, bone mineral density and fat mass.
Muscle fibre characteristics in m. vastus lateralis | Change from baseline to after the training period (10-12 weeks)
  Muscle fiber characteristics such as muscle fiber proportions, cross-sectional area, myonuclei content and capillarization measured in biopsies from m. vastus lateralis
Total-RNA abundance in m. vastus lateralis | Change from baseline to after the training period (10-12 weeks)
  Total-RNA abundance measured in biopsies from m. vastus lateralis.
Total-RNA abundance in m. vastus lateralis | Change from baseline to after 6 training sessions
  Total-RNA abundance measured in biopsies from m. vastus lateralis.
rRNA/RNA abundances in m. vastus lateralis | Change from baseline to after the training period (10-12 weeks)
  rRNA/RNA abundances measured in biopsies from m. vastus lateralis.
rRNA/mRNA abundances in m. vastus lateralis | Change from baseline to after 6 training sessions
  rRNA/RNA abundances measured in biopsies from m. vastus lateralis.
Protein abundances in m. vastus lateralis | Change from baseline to after the training period (10-12 weeks)
  Protein abundances measured in biopsies from m. vastus lateralis.
Protein abundance in m. vastus lateralis | Change from baseline to after 6 training sessions
  Protein abundances measured in biopsies from m. vastus lateralis.
rDNA content in m. vastus lateralis | Measured at baseline
  Ribosomal DNA content measured in m. vastus lateralis
rDNA content in m. vastus lateralis | Change from baseline to after the training period (10-12 weeks)
  Ribosomal DNA content measured in m. vastus lateralis
rDNA content in m. vastus lateralis, (mid) | Change from baseline to after 12 sessions
  Ribosomal DNA content measured in m. vastus lateralis
rDNA content, whole-blood | Measured at baseline
  Ribosomal DNA content measured in whole-blood
rDNA content, whole-blood | Change from baseline to after the training period (10-12 weeks)
  Ribosomal DNA content measured in whole-blood
rDNA content, whole-blood (mid) | Change from baseline to after 12 sessions
  Ribosomal DNA content measured in whole-blood
Epigenetic traits, muscle | Measured at baseline
  Epigenetic traits measured as DNA methylation/histone modifications in m. vastus lateralis
Epigenetic traits, muscle | Change from baseline to after the training period (10-12 weeks)
  Epigenetic traits measured as DNA methylation/histone modifications in m. vastus lateralis
Epigenetic traits, muscle | Change from baseline to after 12 sessions
  Epigenetic traits measured as DNA methylation/histone modifications in m. vastus lateralis
Blood pressure | Change from baseline to after the training period (10-12 weeks).
  Resting blood pressure
Hemoglobin mass | Change from baseline to after the training period (10-12 weeks).
  Total hemoglobin mass measured using the carbon monoxide rebreathing method
Glucose tolerance | Change from baseline to after the training period (10-12 weeks).
  Blood glucose and endocrine responses to a 2h glucose tolerance test (75 g bolus of glucose).
Systemic inflammation | Change from baseline to after the training period (10-12 weeks).
  Systemic inflammation measured as blood markers such as C-reactive protein (CRP) in resting blood samples.
Lipoproteins and lipids in blood | Change from baseline to after the training period (10-12 weeks)
  Concentrations of various lipoproteins and lipids in blood measured using targeted metabolomics
Hemoglobin glycosylation | Change from baseline to after the training period (10-12 weeks)
  Long-term glucose levels measured as hemoglobin glycosylation
Hormone concentrations in blood | Change from baseline to after the training period (10-12 weeks)
  Concentrations of hormones such as testosterone, growth hormone, thyroid hormones, cortisol and insulin (c-peptide) in serum
Health-related quality of life (SF-36) | Change from baseline to after the training period (10-12 weeks)
  Health-related quality of life measured using the SF-36 questionnaire
SARC-F | Measured at baseline
  Sarcopenia score assessed using SARC-F (questionnaire)
SARC-F | Change from baseline to after the training period (10-12 weeks)
  Sarcopenia score assessed using SARC-F (questionnaire)
Dietary registration | Measured at baseline
  Dietary composition assessed using a food-frequency questionnaire (nutritional composition, energy intake, habitual patterns of dietary intake)
Dietary registration | Measured after 12 sessions
  Dietary composition assessed using a food-frequency questionnaire (nutritional composition, energy intake, habitual patterns of dietary intake)
Training diary relating to the intervention protocol | Throughout the intervention (continuous)
  Information about intervention-specific training, including training frequency, volume and load
Activities of daily living (questionnaire) | Measured at baseline
  Activities of daily living measured using a questionnaire (i.e. time spent in activity, intensities and type of activity)
Daily activity level | Measured during the intervention
  Daily activity level registred over three to five days using an accelerometer.

CONTACTS AND LOCATIONS:
Overall Officials: Stian Ellefsen, PhD, Principal Investigator — Inland Norway University of Applied Sciences
Locations (1):
- Inland Norway University of Applied Sciences, Lillehammer, Norway

IPD SHARING:
Plan to Share IPD: Yes
The full data sets used to analyze study outcomes will be made available with the publication of the study. Data sets will be included or referred to in the publication and hosted online.
Supporting Information: Study Protocol, Analytic Code